CLINICAL TRIAL: NCT06793046
Title: Comparisons of Phasic and Terminal Detrusor Overactivity in Women with Lower Urinary Tract Dysfunction
Brief Title: Comparisons of Phasic and Terminal DO
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Principal Investigator, National Taiwan University Clinical Trial Center, Ho-Hsiung Lin, Department of Obstetrics and Gynecology, Principal Investigator, Professor, National Taiwan University Hospital
Other Study IDs: 202406143RINE
Record Dates: First submitted 2025-01-14; First posted 2025-01-27 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2024-07

CONDITIONS: Detrusor Overacitivity
Keywords: Detrusor overactivity
MeSH Terms: conditions — Urinary Bladder, Overactive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Phasic DO: Detrusor involuntary contraction during filling cystometry before strong-desire to void volume
- Terminal DO: Detrusor involuntary contraction at the end of filling cystometry

SUMMARY:
Overactive bladder is a common issue among women of childbearing age, regardless of their childbirth experience. Some of these women may exhibit detrusor overactivity in urodynamic studies. Excluding detrusor overactivity caused by neurogenic bladder, the International Continence Society defines two types of idiopathic detrusor overactivity: phasic and terminal. Although many studies have explored overactive bladder and detrusor overactivity under different conditions, no literature directly compares these two types of detrusor contractions. Therefore, we aim to compare phasic and terminal detrusor overactivity in women with lower urinary tract dysfunction. Between July 2009 and December 2023, medical records of all women with lower urinary tract symptoms who underwent urodynamic studies in the urogynecological department of a medical center were reviewed. The medical records of phasic or terminal detrusor overactivity were selected for comparison (N=290). Those with phasic and terminal detrusor overactivity were excluded (N=21).

DETAILED DESCRIPTION:
Hypothesis / aims of study Detrusor overactivity (DO) can be classified into phasic or terminal ones. However, to our knowledge, clinical and urodynamic differences between phasic or terminal DO have never been reported. Therefore, the objective of this study is to elucidate the above differences.

Study design, materials and methods Between July 2009 and December 2023, medical records, including urodynamic data, bladder dairy data, and questionnaires, including patient perception of bladder condition, urgency severity scale, overactive bladder symptom score, urogenital distress inventory, incontinence impact questionnaire and King's health questionnaire, of all women with lower urinary tract symptoms who underwent urodynamic studies in the urogynecological department of a medical center were reviewed. The medical records of phasic or terminal DO were selected for comparison. Those with phasic and terminal DO were excluded.

STATA software was used for statistical analysis. Wilcoxon rank sum test or chi-square test were used for statistical analysis, as appropriate. A p < 0.05 was considered statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* > 20 y/o
* Women with lower urinary tract symptoms
* Complete urodynamic study with a diagnosis of detrusor overactivity
* Complete the questionnaires

Exclusion Criteria:

* Woman who was pregnant
* Chronic pelvic inflammatory disease

Min Age: 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women more than 20-year-old with lower urinary tract symptoms, received urodynamic study and was diagnosed with detrusor overactivity.
Sampling Method: Non-Probability Sample
Enrollment: 290 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Life quality | Between July 2009 and December 2023
  Use King's health questionnaire Question 2 to evaluate the life quality of the 2 cohort (score 1-4, higher score indicates worse life quality)

SECONDARY OUTCOMES:
Strong-desire to void volume (mL) in urodynamic study | Between July 2009 and December 2023
  Use urodynamic study to evaluate the bladder capacity of the 2 cohort

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Hsiung Lin, M.D. Ph.D, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan, Taiwan

IPD SHARING:
Plan to Share IPD: No
The data will be provided under request.

REFERENCES:
- [Background] Hsiao SM, Wu PC, Chang TC, Chen CH, Lin HH. Urodynamic and Bladder Diary Factors Predict Overactive Bladder-wet in Women: A Comparison With Overactive Bladder-dry. Int Neurourol J. 2019 Mar;23(1):69-74. doi: 10.5213/inj.1836212.106. Epub 2019 Mar 31. PMID 30943696
- [Background] Wu PC, Hsiao SM, Lin HH. Prevalence and predictors of nocturnal polyuria in females with overactive bladder syndrome. World J Urol. 2022 Feb;40(2):519-527. doi: 10.1007/s00345-021-03865-5. Epub 2021 Nov 11. PMID 34762173
- [Background] Abrams P, Cardozo L, Fall M, Griffiths D, Rosier P, Ulmsten U, Van Kerrebroeck P, Victor A, Wein A; Standardisation Sub-Committee of the International Continence Society. The standardisation of terminology in lower urinary tract function: report from the standardisation sub-committee of the International Continence Society. Urology. 2003 Jan;61(1):37-49. doi: 10.1016/s0090-4295(02)02243-4. No abstract available. PMID 12559262
- [Background] Aoki Y, Brown HW, Brubaker L, Cornu JN, Daly JO, Cartwright R. Urinary incontinence in women. Nat Rev Dis Primers. 2017 Jul 6;3:17042. doi: 10.1038/nrdp.2017.42. PMID 28681849
- [Background] Haylen BT, de Ridder D, Freeman RM, Swift SE, Berghmans B, Lee J, Monga A, Petri E, Rizk DE, Sand PK, Schaer GN; International Urogynecological Association; International Continence Society. An International Urogynecological Association (IUGA)/International Continence Society (ICS) joint report on the terminology for female pelvic floor dysfunction. Neurourol Urodyn. 2010;29(1):4-20. doi: 10.1002/nau.20798. PMID 19941278